CLINICAL TRIAL: NCT01198119
Title: Excision Limits of Oral Cavity Tumor by NARROW BAND IMAGING (NBI): Feasibility Trial
Brief Title: Excision Limits of Oral Cavity Tumor by Narrow Band Imaging
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NBI-CAB-0907
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Cancer
Keywords: oral cavity tumor; narrow band imaging; subclinical cancer lesion
MeSH Terms: conditions — Neoplasms; Mouth Neoplasms | interventions — Biopsy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with oral cavity cancer (Experimental): Patient treated by surgery for the oral cavity cancer
  Interventions: Device: Location of the suspected lesions; Procedure: Biopsy; Procedure: Lesion excision/Surgery

INTERVENTIONS:
Device: Location of the suspected lesions — The suspected lesions will be located before the excision, during the surgery.
  1. With traditional light
  2. NBI technique The images will be recorded and compared
Procedure: Biopsy — In case of suspected lesions detected by the NBI technique, this area is biopsied
Procedure: Lesion excision/Surgery — In case of positive biopsy, the suspected lesions is excised

SUMMARY:
This study evaluates the feasibility of the NBI technique in the detection of early cancer lesions.

ELIGIBILITY:
Inclusion Criteria:

* Primitive epidermoid cancer of the oral cavity, proved by histology, not treated previously, patient having a surgery
* No previous surgery for this cancer
* Age > 18 years
* Patient affiliated to health insurance
* Consent signed by the patient

Exclusion Criteria:

* Metastatic or recurrent disease
* Health care impossibilities for geographic, social, psychic reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-07; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Reliability for detection of subclinical lesions | baseline
  Concordance between the histological data and the lesions detected by the NBI technique

SECONDARY OUTCOMES:
Excision limits quality criteria | baseline
  percentage of detection / percentage of false-negative
Detection of suspect lesions | baseline
  Identify the detection of suspect lesions, aloof from the primitive lesion (percentage of detection / percentage of true-positive)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie EL BEDOUI, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France